CLINICAL TRIAL: NCT03665545
Title: Pembrolizumab in Association With the Multipeptide Vaccine IMA950 Adjuvanted With Poly-ICLC for Relapsing Glioblastoma: a Randomized Phase I/ II Trial
Brief Title: Pembrolizumab in Association With the IMA950/Poly-ICLC for Relapsing Glioblastoma
Acronym: IMA950-106
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Denis Migliorini, Principal Investigator, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMA950-106/CER 2018-00718; MK3475-480 (Other: MSD)
Record Dates: First submitted 2018-09-01; First posted 2018-09-11 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Glioblastoma Multiforme; Glioblastoma, Adult; Glioma of Brain; Glioblastoma Multiforme of Brain
Keywords: glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IMA950/Poly-ICLC (Active Comparator): IMA950 mixed with Poly-ICLC administered subcutaneously
  Interventions: Drug: IMA950/Poly-ICLC
- IMA950/Poly-ICLC and pembrolizumab (Experimental): Pembrolizumab 200mg q3w IV and IMA950 mixed with Poly- ICLC administered subcutaneously
  Interventions: Drug: IMA950/Poly-ICLC; Drug: IMA950/Poly-ICLC and pembrolizumab

INTERVENTIONS:
Drug: IMA950/Poly-ICLC — IMA950 mixed with Poly-ICLC administered subcutaneously
Drug: IMA950/Poly-ICLC and pembrolizumab — IMA950 mixed with Poly-ICLC administered subcutaneously in combination with pembrolizumab
  Arms: IMA950/Poly-ICLC and pembrolizumab

SUMMARY:
Monocentric randomized phase I/II trial, including 24 patients diagnosed with relapsing glioblastoma (GBM) irrespective of MGMT and IDH gene status.

Following diagnosis of relapsing glioblastoma by either brain CT scan or MRI, patients will be randomized in 2 arms:

1. Arm 1: IMA950 mixed with Poly-ICLC administered subcutaneously
2. Arm 2: Pembrolizumab 200mg q3w IV and IMA950 mixed with Poly-ICLC administered subcutaneously

The first phase of treatment will last 6 weeks, then surgery will be performed (done if clinically possible ad indicated). In case of available brain tissue, extensive analysis of the tumor immune response will be performed. Assessment of systemic immune response by PBMC immunomonitoring will be systematically done before and after surgery.

DETAILED DESCRIPTION:
Brain tumors are the first cause of cancer mortality in children and the 3rd cause in young adults. The most frequent brain tumors are gliomas and among them the most common type is astrocytoma. The most malignant astrocytoma is Glioblastoma (GBM). Standard therapy of newly diagnosed GBM patients includes surgery, irradiation and temozolomide (TMZ) chemotherapy with 1-year and 5-year survival rates at 30% and 3%, respectively. For the treatment of recurrent GBM, TMZ is widely used even if the optimal dosing schedule and the minimal time interval from first line are unknown. Other appropriate therapeutic options include Lomustine, an alkylating drug, and Bevacizumab, an anti-angiogenic agent targeting VEGF-A, approved only in selected countries (i.e. North America, Switzerland). Controlled trials are rare for recurrent glioblastoma, consequently therapeutic decisions are mostly based on low-level evidence.

Amongst innovative strategies, immunotherapy is considered as one of the most promising. Immunotherapy stimulates the natural properties of the immune system to protect against cancer growth. Therapeutic vaccines (active immunotherapy) are expected to elicit a cytotoxic immune response to tumor-associated antigens, destroying malignant cells without harming normal cells. The cells involved in this response are T lymphocytes, which can sense abnormal peptides at the tumor cells surface. One critical step towards the development of therapeutic vaccines was the identification and validation of glioma antigens. This is an obstacle the investigators have circumvented with the characterization of several immunogenic glioma peptides by screening the peptidome of ex vivo human glioma samples. This led to the development of a multipeptide vaccine called IMA950.

IMA950 is composed of 9 synthetic tumor-associated HLA-A2-restricted peptides (TUMAPs), two MHC class II-binding peptides and one HLA-A2-restricted HBV-derived peptide, the latter used as marker of vaccine immunogenicity. The HLA-A2 allele is expressed by approximately 45% of the Swiss population. As the interactions between peptides and their corresponding HLA molecule are highly specific, only HLA-A*02 positive patients will be included in this trial. The reasons why this set of peptides is very promising for vaccination are as follows:

1. Tumor peptides have been isolated from ex vivo samples:
2. They are over-expressed in glioma (compared to normal tissues)
3. They are derived from proteins involved in the malignant process
4. They are immunogenic in vitro in healthy donors and in glioma patients
5. This is a MULTI-peptide vaccine IMA950 was investigated in a monocentric phase I/II trial for newly diagnosed glioblastoma and WHO grade III gliomas using poly-ICLC as adjuvant (PI: P-Y. Dietrich, NCT01920191, study completed, final results in preparation for publication). A total of 19 patients (16 with GBM and 3 with anaplastic astrocytoma) were included, with a median number of 9 injections received per patient (range: 4-11). The multipeptide vaccine did not show any serious safety issues, apart from some mild inflammatory reactions at the injection site, peritumoral or resection cavity edema/tumor flare manageable with steroids, as well as peri-vaccinational transient mild headache, fatigue and flu-like syndrome (grade 3 events: 42.1%, grade 4 events: 21%, no grade 5 events). Regarding vaccine immunogenicity, CD4 T-cell responses were detected in the majority of patients (58%) and were usually sustained. The CD8 T-cell responses were detected in 63% of patients, with 37% of them being multi-TUMAP responders. Median overall survival from date of surgery was 21 months (range: 10 - 41 months) for the overall cohort, with a 19 months survival for the GBM-only cohort (range: 10-41 months), which compares favorably with the reported median survival of 15 months with the reference treatment of temozolomide-based chemoradiation. PFS was 93% and 56% at 6 and 9 months respectively.

Despite the T cell ability to detect tumor peptides that are naturally presented by tumor cells, these T cells do not normally become activated and do not protect the body against the cancer, as tumor cells on their own are only poorly immunogenic. For effective T cell activation, the help of co-stimulatory molecules, which are expressed on activated professional APCs, e.g. dendritic cells, is required. During infections, the activation of APCs is triggered by molecular patterns common to all pathogens of a class (e.g. RNA viruses). These patterns, also referred to as "danger signals", are not provided by peptides themselves. Consequently, artificial danger signals have to be provided with a tumor vaccine to induce the required co-stimulation on APCs. In combination with a vaccine, such substances with a non-specific immunostimulatory effect are called adjuvants. Poly-ICLC, (Hiltonol®, Oncovir) is a synthetic double-stranded ribo-nucleic acid (dsRNA) mimicking viral pathogen associated molecular patterns (PAMP) that activates multiple elements of innate and adaptive immunity.

The importance of intact immune surveillance in controlling outgrowth of neoplastic cells has been known for decades. The PD-1 receptor-ligand interaction is a major pathway hijacked by tumors to suppress immune control. The normal function of PD-1, expressed on the cell surface of activated T-cells under healthy conditions, is to down-regulate unwanted or excessive immune responses, including autoimmune reactions. Binding of PD-1 ligands (PD-L1 and PD-L2) to the PD-1 receptor inhibits T-cell activation triggered through the T-cell receptor. Pembrolizumab (Keytruda™) is a potent and highly selective humanized monoclonal antibody (mAb) designed to directly block the interaction between PD-1 and its ligands. Impressive response rate and prolonged survival were first observed for metastatic melanoma, but the clinical benefit of this mAb was recently shown to extend to several other cancer types. There is a strong rationale to investigate the role of PD-1/PD-L1 blockade in malignant glioma, since (i) we and others have previously reported that PD-L1 expression by glioma cells may contribute to tumor-related immunoresistance; (ii) PD-L1 is also expressed by tumor-infiltrating macrophages and circulating monocytes; (iii) expression of PD-L1 on circulating monocytes was shown to correlate with worsened survival in patients who received the HSPPC-96 vaccine for newly diagnosed and recurrent GBM. The 200 mg Q3W dose will maintain individual patient exposures within the exposure range demonstrated to be well tolerated, safe and established in melanoma as associated with maximal efficacy response. A fixed dose regimen simplifies the dosing regimen so as to be more convenient for physicians and to reduce the potential for dosing errors.

The combination of pembrolizumab with a vaccine therapy is currently being tested in several trials for different tumors, such as melanoma, bladder, colorectal and prostate cancer (NCT02574533, NCT02054520, NCT02432963, NCT02499835, NCT02515227). Here the investigators postulate that Pembrolizumab may improve the immunogenicity of the IMA950 vaccine and the function of vaccine-induced glioma-specific T cells, and that the multipeptide vaccine may help to focus the immune response against antigens overexpressed by glioma, leading together to an optimization of the antitumor immune effect whilst reducing the risk of collateral damage to the brain.

The study aims to answer questions regarding safety (for the future clinical development of this strategy), immunogenicity (synergy between multipeptide vaccine and pembrolizumab) and clinical outcome. Ancillary translational research should help to identify possible correlation between neo-epitopes, methylation status, immune response and clinical outcome.

ELIGIBILITY:
1. Histological documentation of glioblastoma (de novo or secondary GBM).
2. Patient must be at first or subsequent relapse.
3. HLA-A*0201 positive patients (after pre-screening).
4. ECOG performance status of 0 or 1.
5. Age > 18 years, life expectancy of least 4 months.
6. Patient must be on stable or decreasing dose of steroids administered for glioblastoma, with a maximal dose of Dexamethasone of 4mg/day or equivalent.
7. Adequate bone marrow, liver and kidney function (see Table 2 for definition).
8. Negative Hepatitis B serology (HBcAg-seronegative).
9. Capable of co-operating with the protocol schedule of Pembrolizumab combined with IMA950 and Poly-ICLC and follow-up.
10. Have measurable disease according to the iRANO criteria. Tumor lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
11. Be willing and able to provide written informed consent for the trial.
12. Be willing to provide tissue from a study-specific biopsy of a tumor lesion.
13. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. A urine test can be considered if the serum test is not available.
14. Female subjects of childbearing potential (Section 5.6.2) must be willing to use 2 methods of contraception or be surgically sterile, or abstain from heterosexual activity as outlined in Section 5.6.2 - Contraception, for the course of the study through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been in menopause for more than one year.

    Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
15. Male subjects of childbearing potential must agree to use an adequate method of contraception as outlined in Section 5.6.2- Contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

5.1.4. Main Study Exclusion Criteria

The subject must be excluded from participating in the trial if the subject:

1. Any other vaccination given within 2 weeks before first IMA950 vaccination.
2. Diagnosis of immunodeficiency or active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a condition other than glioblastoma that requires systemic steroids (> 10mg/day prednisone or equivalent) or immunosuppressive agents. Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
3. Patients with evidence of history bleeding diathesis.
4. Pregnant or breastfeeding patients, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
5. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
6. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
7. Has a known history of active TB (Bacillus Tuberculosis)
8. Hypersensitivity to pembrolizumab or any of its excipients.
9. Has had a prior anti-cancer monoclonal antibody within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
10. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

    Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.

    Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
11. Has known history of, or any evidence of active (non-infectious) pneumonitis that required(s) steroids.
12. Has an active infection requiring systemic therapy.
13. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
14. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
15. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
16. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
17. Has known past or active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected). Only patients with negative serology for past or current exposure to HBV and HCV will be eligible.
18. Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however, intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-10-25 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-04-24 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | From the time of treatment randomization through 30 days following cessation of treatment
  To assess tolerability and safety of IMA950 adjuvanted with Poly-ICLC when given together with pembrolizumab, using CTCAE v.4.03

SECONDARY OUTCOMES:
Progression-free survival at 6, 9, 12 months | through study completion, an average of 3 years
  To estimate 6, 9 and 12-month progression-free survival (PFS) using gadolinium-enhanced MRI and clinical assessment according to revised iRANO criteria
Overall Survival | through study completion, an average of 3 years
  To estimate OS, defined as the time between the date of study entry and the date of death due to any cause. Subjects who have not died at the time of last known follow-up will be censored
Patient-reported Quality of life | through study completion, an average of 3 years
  Quality of life patient-reported outcomes (EORTC QLQ-C30 questionnaire)

OTHER OUTCOMES:
Tumor Infiltrating Lymphocyte (TIL) density | through study completion, an average of 3 years
  To assess synergy/immunogenicity of IMA950 plus Poly-ICLC when given together with Pembrolizumab using Tumor Infiltrating Lymphocyte (TIL) density assessment
Vaccine-specific CD4 and CD8 cells | through study completion, an average of 3 years
  To assess synergy/immunogenicity of IMA950 plus Poly-ICLC when given together with Pembrolizumab by assessing vaccine-induced peripheral immune responses by flow cytometry or IHC as surrogate markers

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Mach, Prof., Study Director — University Hospital, Geneva
Locations (1):
- University Hospitals of Geneva, Geneva, Switzerland